CLINICAL TRIAL: NCT05155501
Title: Clinical TrIAL of Approaches to Prostate cAncer suRgery
Acronym: PARTIAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-07023781; 1R01CA259173 (NIH)
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: radical prostatectomy; nerve sparing; Retzius sparing
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors (i.e., pathologists) will be blinded to randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted radical prostatectomy (RP) (Active Comparator): The conventional robotic-assisted radical prostatectomy is the gold standard approach to prostate cancer surgery.
  Interventions: Procedure: Robot-assisted radical prostatectomy (RP)
- Pelvic fascia-sparing robot-assisted radical prostatectomy (PFS-RP) (Experimental): A novel, posterior approach to radical prostatectomy that preserves the dorsal vascular complex, nerves and fascial support structures that overlie the anterior prostate. These structures are disrupted and removed during conventional radical prostatectomy.
  Interventions: Procedure: Pelvic fascia-sparing robot-assisted radical prostatectomy (PFS-RP)

INTERVENTIONS:
Procedure: Robot-assisted radical prostatectomy (RP) — The conventional approach to prostate cancer surgery
  Arms: Robot-assisted radical prostatectomy (RP)
Procedure: Pelvic fascia-sparing robot-assisted radical prostatectomy (PFS-RP) — A novel, posterior approach to radical prostatectomy that preserves the dorsal vascular complex, nerves and fascial support structures that overlie the anterior prostate.
  Arms: Pelvic fascia-sparing robot-assisted radical prostatectomy (PFS-RP)

SUMMARY:
This is a prospective, randomized controlled trial to compare cancer control and health-related quality of life following pelvic fascia-sparing radical prostatectomy versus standard radical prostatectomy.

The investigators hypothesize that pelvic fascia-sparing radical prostatectomy will have similar cancer control (primary outcome) and sexual function outcomes; and significantly better urinary function, penile shortening/deformity and inguinal hernia risks as compared to radical prostatectomy.

DETAILED DESCRIPTION:
Traditional radical prostatectomy is the most popular treatment for clinically significant prostate cancer, however significant risks including urinary incontinence, erectile dysfunction, penile shortening, penile curvature/ deformation (Peyronie's disease), and inguinal hernia, are common. Pelvic fascia-sparing radical prostatectomy is a new surgical technique that may preserve fascial support structures, arterial supply to the penis, and nerves that are severed and resected during conventional radical prostatectomy.

This study will enroll adult men undergoing radical prostatectomy for clinically localized prostate cancer. Subjects will be randomized to receive either radical prostatectomy or pelvic fascia-sparing radical prostatectomy. Investigators will compare cancer control and health-related quality of life outcomes through patient questionnaires and medical record review.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age ≥40 years or ≤80 years
* Scheduled for radical prostatectomy for clinically localized prostate cancer
* Able to read and speak English or Spanish
* Willingness to sign informed consent and adhere to the study protocol

Exclusion Criteria:

* Prior major pelvic surgery or radiotherapy
* Suspicion of N1 disease (i.e., any lymph node greater than 1cm in maximal diameter)

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Surgical Margin Status as assessed by surgical pathology results | 1 week post-surgery
  Presence of cancer cells at the prostate margin is standardized as a positive surgical margin through professional guideline consensus.
Biochemical Recurrence as assessed by Prostate Specific Antigen (PSA) | 6 months post-surgery
  Prostate specific antigen (PSA) levels are obtained from standard of care blood tests, and PSA values are measured in ng/mL.
  In accordance with National Comprehensive Cancer Network (NCCN) guidelines, investigators will capture PSA persistence as failure of PSA to fall to undetectable levels, and PSA recurrence as an undetectable PSA after surgery with a subsequent detectable PSA that increases on 2 or more determinations.
Biochemical Recurrence as assessed by Prostate Specific Antigen (PSA) | 12 months post-surgery
  Prostate specific antigen (PSA) levels are obtained from standard of care blood tests, and PSA values are measured in ng/mL.
Biochemical Recurrence as assessed by Prostate Specific Antigen (PSA) | 24 months post-surgery
  Prostate specific antigen (PSA) levels are obtained from standard of care blood tests, and PSA values are measured in ng/mL.

SECONDARY OUTCOMES:
Surgery-Related Adverse Events as assessed by the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to 30 days following surgery
  The questionnaire will include 20 items from the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE), survey items pertinent to short-stay cancer surgery.
  The questionnaire will assess patient-reported complications and adverse events, such as constipation, nausea and vomiting, fever, chills, fatigue, pain, shortness of breath, swelling and bruising, redness and discharge at the surgical incision site, anxiety, and flatulence (ileus). It will also assess patient contacts with physicians and admittance to urgent care or the emergency room.
Change in Urinary and Sexual Function, as measured by the Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP) | Baseline, 1 month, 6 months, 12 months, and 24 months post-surgery
  The Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP) is a 7-item questionnaire assessing two health-related quality of life domains: urinary and sexual function. All questions refer to patients' health and symptoms in the last four weeks.
  Each domain is scored out of 12 points, with higher scores indicating more complications.
  In total, the EPIC-CP score is the final sum of the two domains, with higher scores indicating more issues related to overall prostate cancer quality of life.
Change in Patient-Reported Penile Shortening and Sexual Function, as measured by a 5-item questionnaire | Baseline, 1 month, 6 months, 12 months, and 24 months post-surgery
  This is a 5-item questionnaire, published in the New England Journal of Medicine (NEJM), that has face validity for assessing penile shortening, self-esteem, and erectile function after radical prostatectomy.
  Question 1 assesses patients' perceived penile length post-surgery, compared to penile length at 30 years of age. It consists of two possible responses: Yes or No.
  Questions 2 and 3 assesses patients' ability to obtain and quality of spontaneous morning erections and sexual activity-related erections. It consists of five possible responses: ranging from "No erections" to "Erections always sufficient".
  Question 4 is a visual digital scale assessing patients' present quality of life. It is scored on a scale of 1-7, with higher scores indicating high quality of life.
  Question 5 is a visual digital scale assessing patients' present self-esteem. It is scored on a scale of 1-7, with higher scores indicating high self-esteem.
Change in patient-Reported Penile Curvature/Deformity (Peyronie's Disease), as measured by a 3-item questionnaire | Baseline, 1 month, 6 months, 12 months, and 24 months post-surgery
  This is a validated, 3-item questionnaire assessing presence of Peyronie's disease. The penile deformity items were validated by blinded clinical examination with 100% sensitivity and 99.4% specificity.
  Question 1 assesses penile hardening/plaques in the flaccid state. Question 2 assesses penile curvature in the erect state. Question 3 assesses pain associated with erection. Each question consists of two possible responses: Yes or No.
Patient-reported Decision Regret, as measured by a 5-item questionnaire | 12 months post-surgery
  This is a 5-item questionnaire assessing treatment regret that was developed and validated in men with prostate cancer.
  Each item is scored on a 5 point scale ranging from "Strongly Agree" to "Strongly Disagree". Responses are converted to a score ranging from 0-100, with higher scores indicating more regret.
Patient-reported Decision Regret, as measured by a 5-item questionnaire | 24 months post-surgery
  This is a 5-item questionnaire assessing treatment regret that was developed and validated in men with prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Jim C Hu, MD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (5):
- United States (5):
  - Georgetown University, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - NewYork-Presbyterian Queens, Flushing, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stangl-Kremser J, Kowalczyk K, Schaeffer EM, Allaf M, Scherr D, Yang X, Matoso A, Azumi N, Robinson B, Vickers A, Hu JC. Study protocol for a prospective, multi-centered randomized controlled trial comparing pelvic fascia-sparing radical prostatectomy with conventional robotic-assisted prostatectomy: The PARTIAL trial. Contemp Clin Trials. 2023 May;128:107168. doi: 10.1016/j.cct.2023.107168. Epub 2023 Apr 2. PMID 37015291